CLINICAL TRIAL: NCT05072990
Title: Type 2 Diabetes Mellitus With Obesity and Dyslipidemia Treated by Chinese Herbal Medicine: a Retrospective Study
Brief Title: Type 2 Diabetes Mellitus With Obesity and Dyslipidemia Treated by Chinese Herbal Medicine
Status: Completed | Type: Observational
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Jiaxing Tian, Attending Physician, Department of Endocrinology, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Other Study IDs: 2020-035-KY
Record Dates: First submitted 2021-09-29; First posted 2021-10-11 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes Mellitus in Obese; Dyslipidemia Associated With Type II Diabetes Mellitus
Keywords: type 2 diabetes mellitus; dyslipidemias; obesity; Chinese herbal medicine; retrospective review
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational group
  Interventions: Drug: Chinese herb medicine

INTERVENTIONS:
Drug: Chinese herb medicine — Patients took 200 ml Chinese herb decoction twice a day before breakfast and dinner.

SUMMARY:
This study is a retrospective review of participants who visited Department of Endocrinology, Guang'anmen Hospital and accepted traditional Chinese medicine formula for at least sis months, from January 2015 to December 2020. All the participants should be diagnosed as type 2 diabetes mellitus, obesity and dyslipidemia. Therapeutic effect of traditional Chinese medicine will be evaluated based on the changes of blood glucose, body mass index, blood lipids, and blood pressure.

DETAILED DESCRIPTION:
The diagnostic criteria for type 2 diabetes mellitus and obesity are based on the Guideline for the prevention and treatment of type 2 diabetes mellitus in China (2020 edition). The diagnostic criteria of dyslipidaemia are based on the Chinese Guidelines on Prevention and Treatment of Dyslipidaemia in Adults (2016, revision edition).

ELIGIBILITY:
Inclusion Criteria:

1. Meet at least three of the requirements below; 1) Fasting Plasma Glucose > 6.1 mmol/L or 2-hour Postprandial Blood Glucose > 7.8 mmol/L or diagnosed as type 2 diabetes mellitus; 2) Body Mass Index > 25 kg / m2; 3) Total Cholesterol > 5.2 mmol / L; Or Triglyceride > 1.70 mmol / L; Or Low-Density Lipoprotein > 3.12 mmol / L; Or High-Density Lipoprotein < 1.04 mmol/L. 4) Systolic blood pressure > 130 mmHg or Diastolic blood pressure > 85 mmHg or diagnosed as hypertension;
2. Received 6 months of continuous Chinese herbal medicine treatment;
3. During the period of receiving Chinese herbal medicine, the patients continued to take western medicine according to the doctor's advice as before.
4. During the period of receiving Chinese herbal medicine, diet and exercise continued according to the original routine, and the tests would be reviewed in the same institution.
5. Aged 18 to 80 years at the time of their consent;
6. Signed informed consent.

Exclusion Criteria:

* Patients who had serious heart, lung, liver, kidney and brain diseases; serious infectious or hemorrhagic diseases; serious nervous system diseases, mental instability; or could not cooperate with treatment were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visited Department of Endocrinology, Guang'anmen Hospital, from January 2015 to December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline HbA1c at 3 months, 6 months | 0 month, 3 months, 6 months
Changes from Baseline Fasting Blood Glucose at 3 months, 6 months | 0 month, 3 months, 6 months
Changes from Baseline Low Density Lipoprotein at 3 months, 6 months | 0 month, 3 months, 6 months
Changes from Baseline Triglyceride at 3 months, 6 months | 0 month, 3 months, 6 months
Changes from Baseline Body Mass Index at 3 months, 6 months | 0 month, 3 months, 6 months

SECONDARY OUTCOMES:
Changes from Postprandial Blood Glucose at 6 months | 0 month, 6 months
Changes from Total Cholesterol at 6 months | 0 month, 6 months
Changes from High Density Lipoprotein at 6 months | 0 month, 6 months
Changes from Systolic Blood Pressure at 6 months | 0 month, 6 months
Changes from Diastolic Blood Pressure at 6 months | 0 month, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jiaxing Tian, PhD, Principal Investigator — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (1):
- Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided